CLINICAL TRIAL: NCT00036478
Title: Pilot Study to Evaluate the Use of Phosphorus P31 Nuclear Magnetic Resonance Spectroscopy as a Non-Invasive Means to Evaluate Mitochondrial Dysfunction in HIV-Infected Subjects
Brief Title: Use of Muscle Spectroscopy to Evaluate Mitochondrial Dysfunction in HIV-Infected Patients
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5144; AACTG A5144
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2004-10

CONDITIONS: HIV Infections
Keywords: Pilot Projects; Exercise; Phosphorus Isotopes; Mitochondria; Lactates; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — HIV Infections; Motor Activity

SUMMARY:
The purpose of this study is to see if magnetic resonance spectroscopy (MRS) can be used to detect damage to the mitochondria in HIV-infected patients taking nucleoside reverse transcriptase inhibitor (NRTI) drugs.

HIV-infected patients taking NRTI drugs may have an increase in a chemical in their blood called lactate. High lactate levels may damage the energy source of the cell (mitochondria). Damage to mitochondria may cause lactic acidosis, liver failure, and other problems. It is important to find effective ways to see if the mitochondria of HIV-infected patients have been damaged. This study will see if MRS can be used to determine mitochondrial damage.

DETAILED DESCRIPTION:
NRTI-related mitochondrial toxicity has been implicated in some fatal cases of lactic acidosis and liver failure. In addition, some investigators believe NRTI-related mitochondrial toxicity to be the culprit in the development of peripheral neuropathy and lipodystrophy in HIV-infected patients. There is a need for a sensitive, reproducible, and noninvasive marker of mitochondrial dysfunction. To date, the only available noninvasive marker is lactate, but lactate testing is insensitive and the significance and reproducibility of lactate levels in the HIV-infected population are questionable. Spectroscopy promises to be a very useful alternative for the evaluation of the in vivo effect of NRTIs on mitochondrial function.

Prior to the screening visit, HIV-infected participants must fast for at least 12 hours and refrain from exercise for at least 24 hours. At the screening visit, all participants have blood drawn for lactate measurements and tests for hepatitis B and C. HIV-uninfected participants have an HIV test. Women who are able to become pregnant have a pregnancy test.

Prior to the entry visit, HIV-infected participants must fast for 12 hours and refrain from exercise for 3 days. At the entry visit, all participants have blood drawn for lactate measurements and women have repeat pregnancy tests. Participants have an MRS scan, which takes approximately 60-80 minutes.

ELIGIBILITY:
Inclusion Criteria

Participants in Groups 1 and 2 may be eligible for this study if they:

* Are at least 18 years old.

Participants in Group 1 (HIV-uninfected) may be eligible for this study if they:

* Are HIV-uninfected within 30 days prior to study entry.

Participants in Group 2 (HIV-infected) may be eligible for this study if they:

* Are HIV infected.
* Have been taking an NRTI-containing anti-HIV drug regimen for 8 weeks or more prior to study entry.
* Have a nonexercise venous lactate level greater than 2 times the upper limit of normal (ULN) on 2 repeated measurements.

Exclusion Criteria

Participants in Groups 1 and 2 may not be eligible for this study if they:

* Have severe claustrophobia.
* Have severe symptoms that, in the opinion of the investigator, would interfere with the ability of participants to perform the exercise required for spectroscopy testing.
* Have hepatitis C or B, within 90 days prior to study entry.
* Have taken certain drugs within 30 days prior to study entry.
* Have a medical condition associated with chronic liver disease other than hepatitis C and B.
* Have consumed excessive amounts of alcohol in the past 12 months.
* Are pregnant or breast-feeding.
* Have a foreign object or metal in their body that would impair MRS testing.
* Have or have had peripheral vascular disease.
* Weigh 250 lbs or more.
* Have a family history of mitochondrial disease or have skeletal muscle disease, heart muscle disease, or nervous system conditions without a clearly defined cause that is not related to mitochondria.

Participants in Group 1 (HIV-uninfected) may not be eligible for this study if they:

* Have any active medical condition.
* Use any prescription drugs, except for vitamins or oral contraceptives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, Study Chair
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, La Jolla, California
  - Univ of California, San Diego Antiviral Research Ctr, San Diego, California
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Univ of Nebraska Medical Ctr, Omaha, Nebraska
  - Beth Israel Med Ctr, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee